CLINICAL TRIAL: NCT00764439
Title: Pilot Study on Usage Patterns of a Novel Nicotine Replacement Therapy - A Multi-Center, Open, 3-Week Randomized Low Intervention Study of Two Different Directions for Use in Smokers Motivated to Quit
Brief Title: Pilot Study of a New Nicotine Replacement Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICTDP2010; 2008-002498-11 (EudraCT Number)
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard NRT user direction
  Interventions: Drug: Nicotine replacement therapy
- 2 (Experimental): Novel NRT user direction
  Interventions: Drug: Nicotine replacement therapy

INTERVENTIONS:
Drug: Nicotine replacement therapy — Nicotine replacement therapy with Standard NRT user direction
  Other Names: NRT
  Arms: 1
Drug: Nicotine replacement therapy — Nicotine replacement therapy with a Novel NRT user direction
  Other Names: NRT
  Arms: 2

SUMMARY:
Pilot study of a new nicotine replacement therapy for smoking cessation.

DETAILED DESCRIPTION:
This will be a pilot study of a new nicotine replacement therapy with two different directions for use in smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older male and female cigarette smokers motivated and willing to stop smoking
* female participants of child-bearing potential should use a medically acceptable means of birth control
* evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study and consents to participate

Exclusion Criteria:

* unstable angina pectoris or myocardial infarction during the previous 3 months
* pregnancy, lactation or intended pregnancy (non-pregnancy will be verified by urine pregnancy test for female participants of child-bearing potential)
* participation in other clinical trials within the previous three months and during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Mean hourly and daily number of doses used | throughout study

SECONDARY OUTCOMES:
Mean number of NRT use occasions per day | Week 1, 2, and 3
Ratings of craving/urge to smoke and withdrawal symptoms | Day 1-14, and Day 20
Self-reported continuous abstinence from smoking, verified by an exhaled CO level of less than 10 ppm | Day 1-21
Cotinine levels | At baseline and week 3
Product acceptability | At week 3 visit
Safety Assessments will consist of monitoring and recording all non-serious Adverse Events and Serious Adverse Events , their frequency, severity, seriousness, and relationship to the investigational product. | throughout duration of the study (+ 30 days for spontaneous SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — Global Medical Affairs & Clinical Research, McNeil AB, Sweden
Locations (2):
- United Kingdom (2):
  - Department of Primary Care and General Practice, University of Birmingham, Birmingham
  - Tobacco Dependence Research Centre at Barts and The London Queen Mary's School of Medicine and Dentistry, London